CLINICAL TRIAL: NCT02860780
Title: A Phase 1 Dose-Escalation Study of LY2606368 in Combination With Ralimetinib in Patients With Advanced or Metastatic Cancer
Brief Title: A Study of Prexasertib (LY2606368) in Combination With Ralimetinib in Participants With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16379; I4D-MC-JTJL (Other: Eli Lilly and Company); 2015-005611-33 (EudraCT Number)
Record Dates: First submitted 2016-08-05; First posted 2016-08-09 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2017-11

CONDITIONS: Advanced Cancer; Metastatic Cancer; Colorectal Cancer; Non-small Cell Lung Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — prexasertib; ralimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: prexasertib + ralimetinib (Experimental): Cohort 1: 60 milligrams (mg) prexasertib (LY2606368) given intravenously (IV) and 100 mg ralimetinib given orally.
  Cohort 2: 60 mg prexasertib (LY2606368) given intravenously (IV) and 200 mg ralimetinib given orally.
  Interventions: Drug: prexasertib; Drug: ralimetinib
- Part B1: prexasertib + ralimetinib (colorectal cancer) (Experimental): 60 mg prexasertib (LY2696368) given IV and 200 mg ralimetinib given orally. Participants receive prexasertib IV on Days 1 and 15 and ralimetinib every 12 hours (Q12H) Days 1 and 14 of a 28 day cycle.
  Interventions: Drug: prexasertib; Drug: ralimetinib

INTERVENTIONS:
Drug: prexasertib — Administered IV
  Other Names: LY2606368
Drug: ralimetinib — Administered orally
  Other Names: LY2228820

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug prexasertib in combination with ralimetinib in participants with advanced or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic cancer.
* Able to swallow tablets.
* For Part B, you will need to have colon cancer or non-small cell lung (NSCLC) cancer with KRAS and/or BRAF mutations.
* Discontinued all previous treatments for cancer and recovered from the acute effects from the therapy.

Exclusion Criteria:

* Active infection (fungal, viral, or bacterial).
* Active cancer in your brain or spinal cord.
* Acute or chronic leukemia.
* Serious heart condition.
* Disease that requires immunosuppressant therapy.
* Diagnosis of inflammatory bowel disease.
* Major small bowel resection that interferes with your body's ability to absorb the oral medicine.
* Participated in other clinical trials investigating prexasertib or ralimetinib.
* Pregnant or breastfeeding.
* Other pre-existing conditions or medical history which your doctor will explain to you.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Prexasertib and Ralimetinib | Cycle 1 (28 Days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Prexasertib | Cycle 1 Day 1 through Cycle 3 Day 1 (28 Day Cycles)
PK: Area Under the Curve (AUC) of Prexasertib | Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
PK: Cmax of Ralimetinib | Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
PK: AUC of Ralimetinib | Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
Best Overall Response (BOR): Percentage of Participants with Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), or Not Evaluable (NE) | Baseline to Earliest Objective Progression or Start of New Anticancer Therapy (Estimated up to 32 Weeks)
Disease Control Rate (DCR): Percentage of Participants who Exhibit SD, CR or PR | Baseline through Measured Progressive Disease (Estimated up to 32 Weeks)
Duration of Response (DOR) | Date of CR or PR to Date of Objective Progression or Death Due to Any Cause (Estimated up to 32 Weeks)
Progression Free Survival (PFS) | Baseline to Objective Progression or Death Due to Any Cause (Estimated Up to 32 Weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (2):
  - Carolinas Medical Center, Charlotte, North Carolina
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne, Germany

REFERENCES:
- See also: Click here for more information about this study: A Study of Prexasertib (LY2606368) in Combination With Ralimetinib in Participants With Advanced or Metastatic Cancer — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JTJL#?postal=